CLINICAL TRIAL: NCT06604234
Title: Randomized, Double-blind, Placebo-controlled Study to Evaluate the Impact of the Combination of Three Probiotic Strains on Quality of Life and Symptoms in Peri- and Postmenopausal Women
Brief Title: Impact of a Probiotic Combination on Quality of Life and Symptoms in Peri- and Postmenopausal Women
Acronym: GynMeno
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AB-GynMeno-24
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Menopause
Keywords: Probiotic; Menopause; Quality of life
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): Probiotic formulation comprising Levilactobacillus brevis KABP-052, Lactiplantibacillus plantarum KABP-051 and Pediococcus acidilactici KABP-021
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo comparator arm with identical pharmaceutical form and aspect
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Combination of Levilactobacillus brevis KABP-052, Lactiplantibacillus plantarum KABP-051 and Pediococcus acidilactici KABP-021 in concentration of 1E09 CFU/capsule
  Arms: Probiotic
Other: Placebo — Placebo comparator containing maltodextrin
  Arms: Placebo

SUMMARY:
In this randomized, placebo-controlled, double-blind study, we aim to investigate if the active product consisting of a probiotic blend can improve the quality of life and alleviate symptoms in peri- and postmenopausal women, using validated questionnaires.

DETAILED DESCRIPTION:
Fifty to 80% of women around menopause or already in postmenopause complain about symptoms such as hot flashes, night sweats, sleep disturbances, tiredness, and depression, which negatively impact their quality of life. The aim of this study was to evaluate the effects of a multiprobiotic strain on the quality of life and menopause-associated symptoms. The study is a de-centralized, prospective, randomized, placebo-controlled, double-blind study in which peri- and postmenopausal women will be recruited and randomly assigned (ratio 2:1) to receive either a probiotic blend or placebo formulation in capsules form for 12 weeks. We aim to recruit up to 300 women. On a monthly basis, quality of life will be evaluated by using the validated Spanish Quality of Life Cervantes questionnaire. In addition, other questionnaires will be administered to monitor menopause-related symptoms (Menopause Rating Scale, MRS) and health-related quality of life (Utian Quality of Life). This will be documented through a specifically designed, web-based platform. Main study variable is change in the global score in MRS scores and Cervantes quality of life scores throughout study period.

ELIGIBILITY:
Inclusion Criteria:

1. Women in peri- and/or postmenopause period (up to 5 years after last menstruation) Perimenopause is defined as if changes in the menstrual cycle (such as longer or shorter cycles, absence of any menstrual cycle, or abnormally heavy or prolonged bleeding) have occurred in the previous 12 months.
2. Age 45-60 years.
3. Cervantes quality of life scale score ≥ 38 at the screening visit.
4. Willing to sign the informed consent.
5. Willing to maintain dietary or lifestyle habits during the study.

Exclusion Criteria:

1. Regular use of probiotics other than the probiotics under study (in the form of food supplements or in foods such as "bifidus" type yogurt) in the month prior to the baseline visit.
2. Use of oral or injectable antibiotics in the last month before the start of the study.
3. Women with history of hysterectomy (removal of the uterus) or ovariectomy (removal of the ovaries).
4. Diagnosis of active oncological disease.
5. Use of hormone replacement therapy (HRT), hormonal analogues or oral contraceptives in the 3 months prior to the start of the study.
6. Type 1 diabetes.
7. Untreated or unstable thyroid disease.
8. Diagnosis of severe renal, cardiac or hepatic disease.
9. Diagnosis of chronic gastrointestinal disease: inflammatory bowel disease (Crohns disease, ulcerative colitis), pancreatitis, short bowel syndrome.
10. Diagnosis of celiac disease
11. Regular intake of laxatives such as polyethylene glycol or irritant laxatives (bisacodyl, sennosides, sodium pyrosulphate) (+3 days/week).
12. Primary or secondary immunodeficiency: AIDS, immunoglobulin deficiency.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 245 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Quality of life measured by the Cervantes Scale | Baseline, 30 days, 60 days, 90 days
  Changes in the Cervantes Scale T standardized score obtained using the mean and standard deviation of the population of young women (20-44 years). Cervantes scale is a validated questionnaire developed for Spanish population comprising 31 items which score from 0 to 5
Menopause-related symptoms evaluated by Menopause Rating Scale (MRS) scale | Baseline, 30 days, 60 days, 90 days
  Changes in total MRS score throughout the study. MRS is a 11-item validated questionnaire, each item scoring from 0 to 4. Scores ranging from 0-4, 5-8, 9-15, and 16+ are used to rate the perceived symptoms as none/minimal, mild, moderate, and severe, respectively

SECONDARY OUTCOMES:
Quality of life measured by the Cervantes Scale subscores | Baseline, 30 days, 60 days, 90 days
  Changes in the subscores of the different domains of the Cervantes® Scale: Menopause and Health, Psychological, Sexuality and Relationship.
Menopause-related symptoms evaluated by MRS scale sub-scores | Baseline, 30 days, 60 days, 90 days
  Changes in the subscores of the different domains of the MRS Scale: Vegetative, Urogenital and Mental.
Utian Quality of Life scale | Baseline, 90 days
  Changes in quality of life total score and sub-scores using the Utian Quality of Life (UQOL) scale. This scale measures quality of life in perimenopause period and comprises 23 items evaluating the following domains: occupational, health, emotional and sexual QOL
Gastrointestinal symptoms | Baseline, 90 days
  Assessment of digestive tolerance based on gastrointestinal symptoms documented on the Gastrointestinal Symptom Rating Scale (GSRS).
Symptoms vaginal infections | Baseline, 30 days, 60 days, 90 days
  Number of days with any of the following vaginal symptoms: itching, irritation or abnormal vaginal discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia González Rodríguez, Principal Investigator — HM hospitales
Locations (1):
- HM Gabinete Velázquez, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Honda S, Tominaga Y, Espadaler-Mazo J, Huedo P, Aguilo M, Perez M, Ueda T, Sawashita J. Supplementation with a Probiotic Formula Having beta-Glucuronidase Activity Modulates Serum Estrogen Levels in Healthy Peri- and Postmenopausal Women. J Med Food. 2024 Aug;27(8):720-727. doi: 10.1089/jmf.2023.k.0320. Epub 2024 Jun 16. PMID 38742994